CLINICAL TRIAL: NCT00832455
Title: A 12 Week Multicenter, Open-label, Observational Study to Evaluate the Effectiveness of Montelukast Sodium (Singulair®), 4 or 5 mg/Day in Pediatric Subjects With Uncontrolled Asthma
Brief Title: Pediatric ACTION3 (Identify, Treat, Control): Effectiveness of Adding Montelukast in Pediatric Subjects With Uncontrolled Asthma (0476-385)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-385; MK0476-385; 2009_523
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2010-02-05 (Estimated); Last update posted 2024-05-13 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Single Person

ARMS (1):
- Montelukast (Experimental)
  Interventions: Drug: montelukast sodium

INTERVENTIONS:
Drug: montelukast sodium — Montelukast 4-5 mg for 12 weeks, oral tablet
  Other Names: Singular

SUMMARY:
a study to describe patient and physician satisfaction with montelukast therapy for the control of asthma used either as monotherapy or in combination with inhaled corticosteroids

ELIGIBILITY:
Inclusion Criteria:

* Patient Is Diagnosed With Asthma For At Least 6 Months
* Patient's Peak Expiratory Flow (PEF) Is 80% Of Predicted Value (Appendix 10)
* Patient Is Currently Untreated, Or Patient Is A User Of Short-Acting 2-Agonist On An As-Needed Basis, Or Patient Is A User Of Ics At Any Dosage
* Physician And/Or Patient Are Dissatisfied With Current Controller Therapy, Or Patient Is Reluctant To Take Ics Therapy, Or Patient Is Insufficiently Controlled Due To Non-Adherence With Current Therapy Through The Preceding 6 Weeks

Exclusion Criteria:

* As Per Canadian Guidelines, Patient Is On A Laba Alone (Formoterol (Oxeze), Salmeterol (Serevent)) Or A Combination Product (Advair Or Symbicort)
* Patient Is Well Controlled, Adherent And Satisfied With Current Controller Therapy

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 445 (Actual)
Dates: Start 2006-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berube D, Djandji M, Sampalis JS, Becker A. Effectiveness of montelukast administered as monotherapy or in combination with inhaled corticosteroid in pediatric patients with uncontrolled asthma: a prospective cohort study. Allergy Asthma Clin Immunol. 2014 May 6;10(1):21. doi: 10.1186/1710-1492-10-21. eCollection 2014. PMID 24932181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: JUN-19-2006
  Last patient out: OCT-28-2008
  Total number of sites: 37 sites in Canada
Groups:
- Montelukast: Montelukast 4-5 mg for 12 weeks, oral tablet
Period: Overall Study
Arm/Group | Montelukast
Started | 445 (445 - number of patients that signed the informed consent form (Safety population))
Baseline | 420 (420 -patients that received at least one dose of study medication and had 1 follow-up visit (ITT))
Week 4 | 411
Week 8 (Optional) | 247
Week 12 | 373
Completed | 373
Not Completed | 72
Not completed — Adverse Event | 13
Not completed — Lost to Follow-up | 26
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 17
Not completed — Screening Failure | 2
Not completed — Stopped Medication | 4
Not completed — Parent misunderstood study | 1
Not completed — Parent dissatisfied | 1
Not completed — No improvement | 3
Not completed — Patient moved | 1

BASELINE CHARACTERISTICS:
Arm/Group | Montelukast
Number analyzed (Participants) | 420
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.00 (3.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168
  Male | 252
ICS (Inhaled Corticosteroids) Use [Number; unit: Participants]
  Use | 323
  No Use | 97
Asthma Diagnosis Duration [Mean (Standard Deviation); unit: Months] | 45.58 (34.72)

OUTCOME MEASURES:

1. Primary Outcome: Asthma Control Questionnaire (ACQ)
Description: ACQ is a questionnaire consisting of seven 7-point Likert scale questions describing frequency and severity of asthma symptoms. Score ranges between 0 (well-controlled) and 6 (extremely poorly controlled); a score of ≤0.75 indicates well controlled symptoms.
Time Frame: Week 0, 4, and 12
Population: 420 patients qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit. The following results are based on the 411 patients who completed week 4 and the 373 patients who completed week 12.
Measure: Number; unit: Participants
Groups:
- Montelukast ITT at Week 0; Montelukast ITT at Week 4; Montelukast ITT at Week 12: ITT population, receiving montelukast 4 or 5 mg/day
Arm/Group | Montelukast ITT at Week 0 | Montelukast ITT at Week 4 | Montelukast ITT at Week 12
Number analyzed (Participants) | 420 | 411 | 373
Participants
  Not well controlled | 328 | 159 | 96
  Well controlled | 91 | 251 | 276
  Missing | 1 | 1 | 1
Statistical Analysis 1: Comparison: Montelukast ITT at Week 0 vs Montelukast ITT at Week 12; Test type: Superiority or Other; p < 0.001, McNemar
Statistical Analysis 2: Comparison: Montelukast ITT at Week 0 vs Montelukast ITT at Week 4; Test type: Superiority or Other; p < 0.001, McNemar

2. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: as for outcome 1
Time Frame: Week 0, 4, and 12
Population: 420 patients qualified for inclusion in the intent to treat (ITT) analysis and completed the first visit. The following results are based on the 411 patients who completed week 4, the 247 who completed week 8, and the 373 patients who completed week 12.
Measure: Number; unit: Participants
Arm/Group | Montelukast ITT at Week 0 | Montelukast ITT at Week 4 | Montelukast ITT at Week 12
Number analyzed (Participants) | 420 | 411 | 373
Participants
  Not tapered and Not well controlled | 144 | 60 | 82
  Not tapered and Well controlled | 208 | 121 | 216
  Tapered and Not well controlled | 15 | 14 | 14
  Tapered and Well controlled | 43 | 52 | 60
  Missing | 1 | 0 | 1

3. Other Pre Specified Outcome: Physician Global Satisfaction
Description: At week 0, 4, 8 and 12, physicians were asked to complete a single question describing how satisfied they were regarding the asthma controller medication for each of their enrolled patients.
Time Frame: week 0, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Montelukast ITT at Week 0 | Montelukast ITT at Week 4 | Montelukast ITT at Week 8 | Montelukast ITT at Week 12
Number analyzed (Participants) | 420 | 411 | 247 | 373
Participants
  Very satisfied | 2 | 130 | 116 | 186
  Satisfied | 23 | 148 | 100 | 136
  Neither Satisfied or Dissatisfied | 96 | 101 | 22 | 32
  Dissatisfied | 266 | 28 | 7 | 14
  Very Dissatisfied | 26 | 1 | 0 | 3
  Missing | 7 | 3 | 2 | 2
Statistical Analysis 1: Comparison: Montelukast ITT at Week 0 vs Montelukast ITT at Week 12; Test type: Superiority or Other; p < 0.001, McNemar-Bowker; The McNemar-Bowker test is a statistical procedure used to compare the proportion of physician satisfaction at week 0 compared to week 12
Statistical Analysis 2: Comparison: Montelukast ITT at Week 0 vs Montelukast ITT at Week 8; Test type: Superiority or Other; p < 0.001, McNemar-Bowker; The McNemar-Bowker test is a statistical procedure used to compare the proportion of physician satisfaction at week 0 compared to week 8

4. Other Pre Specified Outcome: Patient Global Satisfaction
Description: At week 0, 4, 8 and 12, patients were asked to complete a single question describing how satisfied they were regarding their asthma controller medication.
Time Frame: Week 0, 4, 8 and 12
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Montelukast ITT at Week 0 | Montelukast ITT at Week 4 | Montelukast ITT at Week 8 | Montelukast ITT at Week 12
Number analyzed (Participants) | 420 | 411 | 247 | 373
Participants
  Very Satisfied | 11 | 145 | 129 | 194
  Satisfied | 62 | 161 | 87 | 120
  Neither Satisfied or Dissatisfied | 137 | 74 | 24 | 48
  Dissatisfied | 190 | 26 | 6 | 7
  Very Dissatisfied | 18 | 3 | 0 | 2
  Missing | 2 | 2 | 1 | 2
Statistical Analysis 1: Comparison: Montelukast ITT at Week 0 vs Montelukast ITT at Week 12; Test type: Superiority or Other; p < 0.001, McNemar-Bowker; The McNemar-Bowker test is a statistical procedure used to compare the proportion of patient satisfaction at week 0 compared to week 12

5. Other Pre Specified Outcome: Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ)
Description: The change in the quality of life of the caregivers of patients treated with montelukast for the control of asthma used in combination with inhaled corticosteroids, using the Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ).
  PACQLQ score ranges between 1 (severe impairment) and 7 (no impairment) where a higher score indicates better quality of life. An average change in overall score ≥0.7 is considered clinically significant. Changes between visits and baseline are described.
Time Frame: Weeks 4, 8, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Montelukast ITT at Week 4 | Montelukast ITT at Week 8 | Montelukast ITT at Week 12
Number analyzed (Participants) | 411 | 247 | 373
Units on a Scale | 1.06 (1.27) | 1.39 (1.39) | 1.36 (1.34)
Statistical Analysis 1: Comparison: Montelukast ITT at Week 12; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Change in PACQLQ score between Week 12 and baseline is statistically different than zero

ADVERSE EVENTS:
Arm/Group | Montelukast
Serious Adverse Events (participants affected / at risk) | 5
Other Adverse Events (participants affected / at risk) | 146
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Montelukast
Bronchitis (Infections and infestations) | 1/445 (1)
Pneumomia (Infections and infestations) | 1/445 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2/445 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1/445 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Montelukast
Pyrexia (General disorders) | 10/445 (10)
Lower respiratory tract infection (Infections and infestations) | 4/445 (4)
Nasopharyngitis (Infections and infestations) | 30/445 (31)
Otitis media (Infections and infestations) | 8/445 (8)
Pharyngitis streptococcal (Infections and infestations) | 4/445 (4)
Pneumonia (Infections and infestations) | 5/445 (5)
Upper respiratory tract infection (Infections and infestations) | 33/445 (33)
Viral infection (Infections and infestations) | 15/445 (15)
Viral upper respiratory tract infection (Infections and infestations) | 4/445 (4)
Headache (Nervous system disorders) | 5/445 (5)
Nightmare (Psychiatric disorders) | 6/445 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 26/445 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 8/445 (8)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4/445 (4)
Rash (Skin and subcutaneous tissue disorders) | 4/445 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.